CLINICAL TRIAL: NCT06295328
Title: From Fungus to Virus, a Phase 1b Clinical Trial Investigating the Safety and Efficacy of Terbinafine in Chronic Hepatitis B Patients
Brief Title: From Fungus to Virus, Investigating the Safety and Efficacy of Terbinafine in Chronic Hepatitis B Patients
Acronym: HepBTer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Ulrich Beuers, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL 72439.018.19
Record Dates: First submitted 2024-02-12; First posted 2024-03-06 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Terbinafine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Phase 1b study with two parallel treatment arms and placebo controls.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- NUC + Study drug (Active Comparator): Tenofovir + Terbinafine
  Interventions: Drug: Terbinafine; Drug: Tenofovir
- NUC + Placebo (Placebo Comparator): Tenofovir + Placebo
  Interventions: Drug: Placebo; Drug: Tenofovir
- Study drug (Active Comparator): Terbinafine
  Interventions: Drug: Terbinafine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Terbinafine — terbinafine 250mg once daily for 4 weeks, followed by 2 weeks washout, followed by 4 weeks bid.
  Arms: NUC + Study drug; Study drug
Drug: Placebo — Placebo 250mg once daily for 4 weeks, followed by 2 weeks washout, followed by 4 weeks bid.
  Arms: NUC + Placebo; Placebo
Drug: Tenofovir — Tenofovir 245mg standard of care
  Arms: NUC + Placebo; NUC + Study drug

SUMMARY:
Rationale: Currently, there is no curative therapy available for patients that are chronically infected with the hepatitis B virus (HBV). Especially the presence of a viral reservoir of stable episomal, covalently closed circular DNA (cccDNA) in the nucleus of infected hepatocytes poses a great challenge for the development of curative therapies. HBV cccDNA acts as the template for production of viral proteins and HBV genomes. In a preclinical study, terbinafine (an antifungal agent) was identified as a potent and specific suppressor of HBx-mediated cccDNA transcription. HBx is an accessory viral protein of HBV which has been proven to be essential for HBV replication and enhances replication at the transcriptional level in vivo. The suppression of cccDNA transcription results in a strong reduction of the production of viral genomes (RNA and DNA) as well as viral proteins. This will allow recovery of the immune system, increase viral clearance and prevent replenishment of the cccDNA pool in the hepatocyte, all contributing to cure chronic hepatitis B (CHB).

Objective: to provide proof of concept for the inhibition of HBx mediated cccDNA transcription by terbinafine, both as monotherapy and add-on therapy next to tenofovir. Secondary outcomes will be the safety and tolerability of terbinafine in this specific group.

Study design: This pilot study is a stratified, single center, randomized, double-blinded, placebo-controlled, dose-ascending proof of concept clinical trial.

Study population: patients chronically infected with the hepatitis B virus with a normal liver function and no signs of liver damage, who do not use any antiviral medication (group A, n=16) or are treated with tenofovir > 6 months (group B, n=16).

Intervention: Patients will be randomly allocated to daily oral treatment with terbinafine or a matched placebo, either as monotherapy (group A) or as add-on therapy to tenofovir (group B).

Main study parameters/endpoints: Primary outcomes: decline in level of serum HBsAg >0.32log10 IU/mL in both groups A and B and decline in serum HBV DNA >0.86log10 in group A at the end of study treatment (week 10 vs baseline). Secondary outcomes: 1) Safety and tolerability of terbinafine as mono- or combination therapy; 2) level of serum HBsAg and HBV DNA at 3 months follow-up; 3) decline of HBsAg levels over time (all visits); 4) HBV RNA, large HBsAg (LHBs) HBcrAg levels, and HBeAg status at baseline and end of study 4).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients participating in this study will undergo physical examinations and blood sample collections (13 samples and in total 467.5 mL). They will also be asked to fill in the HBQOL and EQ5D5L quality of life questionnaires and a medicine diary. In total there will be 13 visits in the hospital of which 7 will be for blood collection only. Terbinafine can induce liver damage 1 of 50,000 to 120,000 prescriptions (LiverTox), a weekly safety laboratory control is implemented in the visits to detect possible liver toxicity in an early stage and prevent liver damage.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60 years
2. Proven CHB for more than 6 months, based on serology (HBsAg positivity) and at screening a viral load of:

   i) Group A: HBV DNA ≥200 IU/mL and <20,000 IU/mL ii) Group B: HBV DNA < 20 IU/mL
3. HBeAg-positive or HBeAg-negative
4. No current use of any antiviral medication (group A) or currently treated with tenofovir only, for > 6 months (group B).
5. Normal liver function tests, assessed as follows:

   i) Liver stiffness measurement using Fibroscan® of ≤ 7.0 kiloPascal (kPa) ii) Alanine aminotransferase (ALT) and/or aspirate aminotransferase (AST) at screening ≤ 1.25 x upper limit of normal (ULN) iii) Thrombocytes 150-400 10E9/L iv) Total bilirubin 0-17 µmol/L (elevated levels may be accepted if unconjugated portion is elevated in patients with Gilbert syndrome) v) Albumin within normal value (35 - 50 g/L) vi) Prothrombin Time (PT) within normal value (9,5 - 12.5 sec) vii) Alkaline phosphatase (ALP) and Gamma-glutamyltransferase (GGT) within normal values (40-120 U/L and 0-40 U/L respectively)
6. Body mass index (BMI): 17.0-35.0 kg/m2
7. Clinical chemistry, hematologic and coagulation tests at screening must be within normal limits or clinically non-significant, as by the investigator's assessment.
8. At screening, women of child bearing potential must be non-pregnant and non-lactating; a urine or serum pregnancy test will be performed at screening.
9. Female patients of child-bearing potential (with a fertile male sexual partner) and male patients (if not surgically sterilized) must be willing to use adequate contraception from screening until last study visit.
10. No recent (<3 months) history of any clinically significant conditions, which, in the opinion of the investigator, would jeopardize the safety of the patient or impact the validity of the study results.
11. Written informed consent must be obtained before any study related interventions (including screening and enrollment) can be conducted.

Exclusion Criteria:

1. Currently active, or a history of liver cirrhosis determined by one or more of the following:

   i) Liver biopsy; ii) Elastography (e.g. Fibroscan); iii) Combination of usual radiological and biochemical criteria
2. Currently active liver disease other than CHB
3. Co-infection with hepatitis C virus (HCV), hepatitis D virus (HDV), hepatitis E virus (HEV) and/or human immunodeficiency virus (HIV)
4. Acute hepatitis A virus (HAV) infection at screening
5. Renal impairment (estimated glomerular filtration rate (eGRF) < 60ml/min)
6. Currently active, or a history of, psoriasis or lupus erythematodes
7. Use of oral medication that interacts with the liver metabolism enzyme CYP2D6, or which is known to be hepatotoxic or otherwise known to interact with terbinafine (such as rifampicin).
8. The use of a L-type calcium (LTCC) blocker (such as lomerizine of nifedipine), since these may interact with the HBV transcription according to the article by Klundert et al.
9. Usage or plans to receive systemic immunosuppressive or immunomodulating medication (e.g. IFN) during the study or ≤4 months prior to the first investigational product administration.
10. Clinical diagnosis of substance abuse ≤12 months prior to screening with narcotics or cocaine or with alcohol (regular consumption >14 units/week [men] and >7 units/week [women])
11. Inability to understand the patient information and make an informed decision to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in level of serum HBsAG | 10 weeks
  - Change in level of serum HBsAg >0.32 log10 IU/mL at the end of study treatment (week 10 vs baseline).
Change in serum HBV DNA | 10 weeks
  - Change in serum HBV DNA >0.86 log10 in group A (monotherapy) at the end of study treatment (week 10 vs baseline).

SECONDARY OUTCOMES:
Safety of terbinafine | 10 weeks
  - Safety of terbinafine as mono- or combination therapy, as defined by the number of patients with treatment-related laboratory adverse events as assessed by CTCAE v4.0.
Tolerability of terbinafine | 10 weeks
  - Tolerability of terbinafine as mono- or combination therapy, as defined by the number of patients with treatment-related adverse events as assessed by CTCAE v4.0
Serum levels of HBsAG | 3 months
  - Level of serum (large) HBsAg at 3 months follow-up.
Serum levels of HBV DNA | 3 months
  - Level of serum HBV DNA at 3 months follow-up.
Serum levels of HBV RNA | 3 months
  - Level of serum HBV RNA at 3 months follow-up.
Serum levels of HBcrAg | 3 months
  - Level of serum HBcrAg at 3 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No